CLINICAL TRIAL: NCT04422054
Title: Correlation Between the Diameter of the Infrarenal Abdominal Aortic Aneurysms Treated With Open or Endovascular Surgical and the Post-procedural Outcomes.
Brief Title: Aneurysm Diameter and Surgical Outcome
Acronym: ADASO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.19.
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Abdominal Aortic Aneurysm; Surgery; Outcome, Fatal
Keywords: open surgery; endovascular repair; aneurysm size; outcome
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Conversion to Open Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open Surgery Repair Group: In the open surgery repair group, preoperative patient characteristics, comorbid conditions, aneurysm anatomy and diameters will be matched with outcomes and complications, in the postoperative period, during follow up.
  Interventions: Procedure: Open Surgery
- Endovascular Repair Group: In the endovascular surgery repair group, preoperative patient characteristics, comorbid conditions, aneurysm anatomy and diameters will be matched with outcomes and complications in the postoperative period, during follow up.
  Interventions: Procedure: Endovascular Surgery

INTERVENTIONS:
Procedure: Open Surgery — We will retrospectively review patients with abdominal aortic aneurysms that underwent open surgical repair.
  Groups: Open Surgery Repair Group
Procedure: Endovascular Surgery — We will retrospectively review patients with abdominal aortic aneurysms that underwent endovascular repair.
  Groups: Endovascular Repair Group

SUMMARY:
Aneurysm diameter is an important risk for rupture and related death in affected patients.

This study will evaluate whether aneurysms size may even influence post procedural outcomes both in open surgical repair and in end-vascular aneurysm repair.

We will retrospectively review clinical data of operated patients with abdominal aortic aneurysm. We will consider both open surgical repair and endovascular aneurysm repair procedures in order to assess the influence of aneurysm size at the time of intervention.

DETAILED DESCRIPTION:
Since the publication by Szilagyi et al, size of aneurysms has been recognized as the predominant risk factor for rupture. In fact, a low risk is associated with small aneurysms, an intermediate risk with medium-sized aneurysms, and dramatically an increased risk with large aneurysms. Current guidelines suggest that the threshold diameter for aneurysm surgery being 5.5 cm for male patients and 5.0 cm for female patients, as measured on the largest section of the aneurysm.

The correlation aneurysm diameter may also have an impact on early and late postoperative outcomes both for open surgery and endovascular surgery. The study by Peppelenbosch N et al. showed that size differences were strongly associated with adverse outcomes during follow-up of patients that underwent endovascular aneurysm repair.

The aim of this is to assess the influence of aneurysm size on the early and late outcomes of open surgical repair (OSR) and endovascular aneurysm repair (EVAR) of abdominal aortic aneurysms (AAA).

Preoperative patient characteristics, comorbid conditions, aneurysm anatomy and diameters will be retrospectively reviewed in order to correlate with the results of the procedures (OSR and EVAR) and with adverse outcome that may have been occurred during follow up.

ELIGIBILITY:
Inclusion Criteria:

* patients with abdominal aortic aneurysm who underwent open surgery or endovascular procedures with complete anatomic data of aneurysms and clinical data with a minimus of 5 years of follow up.

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients, of both sex, with abdominal aortic aneurysm who underwent open surgery or endovascular procedures.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-09-02 (Estimated); Study Completion 2020-10-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between Aneurysm Diameter and Open Surgery Outcome | 5 years of follow up
  We will correlate outcomes and complications with preoperative aneurysm size.
Correlation between Aneurysm Diameter and Endovascular Repair | 5 years of follow up
  We will correlate outcomes and complications with preoperative aneurysm size.

CONTACTS AND LOCATIONS:
Overall Officials: 14743127 Serra, M.D., Ph.D., Principal Investigator — University Magna Graecia of Catanzaro
Locations (1):
- CIFL- Interuniversity Center of Phlebolymphology, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szilagyi DE, Elliott JP, Smith RF. Clinical fate of the patient with asymptomatic abdominal aortic aneurysm and unfit for surgical treatment. Arch Surg. 1972 Apr;104(4):600-6. doi: 10.1001/archsurg.1972.04180040214036. No abstract available. PMID 5013802
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Peppelenbosch N, Buth J, Harris PL, van Marrewijk C, Fransen G; EUROSTAR Collaborators. Diameter of abdominal aortic aneurysm and outcome of endovascular aneurysm repair: does size matter? A report from EUROSTAR. J Vasc Surg. 2004 Feb;39(2):288-97. doi: 10.1016/j.jvs.2003.09.047. PMID 14743127